CLINICAL TRIAL: NCT02922322
Title: Effectiveness of Mat Pilates Exercises in Individuals With Chronic Nonspecific Low Back Pain: A Randomized Controlled Trial
Brief Title: Effectiveness of Mat Pilates Exercises in Individuals With Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Carina Carvalho Correia Coutinho, Adjunct Professor, Head of the Federal University of Paraiba Clinical School of Physical Therapy, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CAAE: 51317315.2.0000.5188
Record Dates: First submitted 2016-06-05; First posted 2016-10-04 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-09

CONDITIONS: Nonspecific Chronic Low Back Pain; Chronic Low Back Pain
Keywords: Mat Pilates; Chronic Nonspecific low back pain; Quality of life; Disability; transverse abdominal muscle

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pilates Group (Active Comparator): The Pilates Group was composed by 15 participants evaluated before and after 16 sessions of intervention with mat Pilates exercises.
  Interventions: Other: Pilates Group
- Control Group (No Intervention): The control group was composed by 15 participants that received no intervention

INTERVENTIONS:
Other: Pilates Group — The Pilates group program (PG) was composed of 16 sessions, 2x per week, 60 minute session each for 8 weeks. The intervention was based on 20 out of the 34 original mat exercises proposed by the Pilates method, classified into basic, intermediate or advanced levels divided into 4 cycles of 5 exercises each. The exercises were performed during two series of 10 repetitions respecting the patients skills.
  Arms: Pilates Group

SUMMARY:
To analyze the effectiveness of mat Pilates compared to no intervention in individuals with chronic nonspecific low back pain.

DETAILED DESCRIPTION:
There is evidence that exercises based on the Pilates method reduce pain in chronic nonspecific low back pain (CNLBP). However, is noticed the lack of studies that compare the effectiveness of mat Pilates to no intervention in the treatment of individual with CNLBP. Therefore, the main objective of the study is to analyze the effectiveness of mat Pilates compared to no intervention in patients with chronic nonspecific low back pain. It is a randomized controlled trial with two arms and double blinded (caregiver, assessor and outcome assessor), composed of 30 patients, aged between 18- 65 years (±22,47) of both sexes, diagnosed with chronic non-specific low back pain persisting for more than three months and pain intensity greater than 3 points in the Pain Numerical Rating Scale. The participants were randomly divided into two groups: Pilates Group (n = 15), intervention based on mat Pilates exercises, and Control Group (n =15) with no intervention. The mat Pilates group performed 16 sessions, twice a week in 60-minute duration each throughout eight weeks, whereas the control group participants kept usual cares until the end of the intervention. Both groups were evaluated before and after the program by a researcher who was unaware of the patients' allocation. The primary assessed outcomes: pain intensity (Pain numerical rating scale, and McGill questionnaire), quality of life (SF-36), and disability (Oswestry Low Back Pain Disability Questionnaire). In addition, the strength and muscle activation of transverse abdominal as secondary outcome assessed through the Stabilizer Pressure Biofeedback Unit test. As a result, the study infers that mat Pilates exercises have significantly improved all the evaluated outcomes. Thus, supporting clinical decisions for the treatment of chronic nonspecific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Complaining of non-specific low back pain for more than three months without radicular symptoms for a period exceeding 12 months.
* Pain intensity equal to or more than 3 points evaluated by the Pain Numerical Rating Scale in the last seven days.
* Eligibility to practice physical activity responding to the Physical Activity Readiness Questionnaire - PAR-Q

Exclusion Criteria:

* Degenerative or inflammatory pathologies of the spine,
* Acute crisis of pain in the shoulders, knees, ankles and spine
* Spinal tumors
* Recent surgery on the spine, lower and upper limbs
* Herniated disc
* Spondylolysis or spondylolisthesis
* Rheumatologic diseases
* Patients who are in labor dispute
* In treatment involving Pilates, physiotherapy or medication.
* Do not understand the writing and speaking Portuguese.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Questionnaire on Pain Intensity | 8 weeks
  The pain intensity was evaluated using an 11-point pain numerical rating scale.

SECONDARY OUTCOMES:
Questionnaire on Quality of Life | 8 weeks
  The quality of life assessment was measured through the SF-36 questionnaire.
Questionnaire on Disability | 8 weeks
  The index of disability was assessed trough the 2.0 version of the Oswestry questionnaire, which is a specific questionnaire to evaluate levels of disability in people who suffer with low back pain.
Questionnaire on Pain Describers | 8 weeks
  The pain describers were evaluated through the MCGill questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: IDEMAR R DOS SANTOS JUNIOR, BPhty, Principal Investigator — Federal University of Paraíba; CARINA CC COUTINHO, MD, Study Director — FEDERAL UNIVERSITY OF PARAIBA

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pereira LM, Obara K, Dias JM, Menacho MO, Guariglia DA, Schiavoni D, Pereira HM, Cardoso JR. Comparing the Pilates method with no exercise or lumbar stabilization for pain and functionality in patients with chronic low back pain: systematic review and meta-analysis. Clin Rehabil. 2012 Jan;26(1):10-20. doi: 10.1177/0269215511411113. Epub 2011 Aug 19. PMID 21856719
- [Background] Hodges PW, Richardson CA. Inefficient muscular stabilization of the lumbar spine associated with low back pain. A motor control evaluation of transversus abdominis. Spine (Phila Pa 1976). 1996 Nov 15;21(22):2640-50. doi: 10.1097/00007632-199611150-00014. PMID 8961451
- [Background] Miyamoto GC, Costa LO, Cabral CM. Efficacy of the Pilates method for pain and disability in patients with chronic nonspecific low back pain: a systematic review with meta-analysis. Braz J Phys Ther. 2013 Nov-Dec;17(6):517-32. doi: 10.1590/S1413-35552012005000127. PMID 24346291
- [Background] Franco YR, Liebano RE, Moura KF, de Oliveira NT, Miyamoto GC, Santos MO, Cabral CM. Efficacy of the addition of interferential current to Pilates method in patients with low back pain: a protocol of a randomized controlled trial. BMC Musculoskelet Disord. 2014 Dec 10;15:420. doi: 10.1186/1471-2474-15-420. PMID 25492853
- [Background] Miyamoto GC, Costa LO, Galvanin T, Cabral CM. The efficacy of the addition of the Pilates method over a minimal intervention in the treatment of chronic nonspecific low back pain: a study protocol of a randomized controlled trial. J Chiropr Med. 2011 Dec;10(4):248-54. doi: 10.1016/j.jcm.2011.06.007. PMID 22654682
- [Background] Kamioka H, Tsutani K, Katsumata Y, Yoshizaki T, Okuizumi H, Okada S, Park SJ, Kitayuguchi J, Abe T, Mutoh Y. Effectiveness of Pilates exercise: A quality evaluation and summary of systematic reviews based on randomized controlled trials. Complement Ther Med. 2016 Apr;25:1-19. doi: 10.1016/j.ctim.2015.12.018. Epub 2016 Jan 4. PMID 27062942
- [Background] La Touche R, Escalante K, Linares MT. Treating non-specific chronic low back pain through the Pilates Method. J Bodyw Mov Ther. 2008 Oct;12(4):364-70. doi: 10.1016/j.jbmt.2007.11.004. Epub 2008 Feb 1. PMID 19083695
- [Background] Rydeard R, Leger A, Smith D. Pilates-based therapeutic exercise: effect on subjects with nonspecific chronic low back pain and functional disability: a randomized controlled trial. J Orthop Sports Phys Ther. 2006 Jul;36(7):472-84. doi: 10.2519/jospt.2006.2144. PMID 16881464
- [Background] Lim EC, Poh RL, Low AY, Wong WP. Effects of Pilates-based exercises on pain and disability in individuals with persistent nonspecific low back pain: a systematic review with meta-analysis. J Orthop Sports Phys Ther. 2011 Feb;41(2):70-80. doi: 10.2519/jospt.2011.3393. Epub 2010 Oct 22. PMID 20972339
- [Background] da Luz MA Jr, Costa LO, Fuhro FF, Manzoni AC, de Oliveira NT, Cabral CM. Effectiveness of mat Pilates or equipment-based Pilates in patients with chronic non-specific low back pain: a protocol of a randomised controlled trial. BMC Musculoskelet Disord. 2013 Jan 9;14:16. doi: 10.1186/1471-2474-14-16. PMID 23298183
- [Background] da Luz MA Jr, Costa LO, Fuhro FF, Manzoni AC, Oliveira NT, Cabral CM. Effectiveness of mat Pilates or equipment-based Pilates exercises in patients with chronic nonspecific low back pain: a randomized controlled trial. Phys Ther. 2014 May;94(5):623-31. doi: 10.2522/ptj.20130277. Epub 2014 Jan 16. PMID 24435105
- [Background] Wajswelner H, Metcalf B, Bennell K. Clinical pilates versus general exercise for chronic low back pain: randomized trial. Med Sci Sports Exerc. 2012 Jul;44(7):1197-205. doi: 10.1249/MSS.0b013e318248f665. PMID 22246216
- [Background] Turner L, Shamseer L, Altman DG, Weeks L, Peters J, Kober T, Dias S, Schulz KF, Plint AC, Moher D. Consolidated standards of reporting trials (CONSORT) and the completeness of reporting of randomised controlled trials (RCTs) published in medical journals. Cochrane Database Syst Rev. 2012 Nov 14;11(11):MR000030. doi: 10.1002/14651858.MR000030.pub2. PMID 23152285